CLINICAL TRIAL: NCT02498340
Title: Diet Challenge in G6PD Deficient Egyptian Children: A One- Year Prospective Single Center Study With Genotype - Phenotype Correlation
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohsen Saleh Elalfy, professor, Ain Shams University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Diet challenge in G6PD
Record Dates: First submitted 2015-07-10; First posted 2015-07-15 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-07

CONDITIONS: Glucose-6-Phosphate Dehydrogenase Deficiency
Keywords: G6PD; genotype; phenotype; diet restriction
MeSH Terms: conditions — Glucosephosphate Dehydrogenase Deficiency

ARMS (1):
- Diet challenge (Experimental): The patients will have a single blood test after dietetic challenge, they will be subjected to eat non- fava beans diet at doses of 10 -30 gm of 3 different types of non- fava beans( each one will be given once daily for 3 days).
  Interventions: Dietary Supplement: non- fava beans

INTERVENTIONS:
Dietary Supplement: non- fava beans — Patients will be subjected to eat non- fava beans diet at doses of 10 -30 gm (small to moderate amount) of 3 different types of non- fava beans, each one will be given once daily for 3 days.

SUMMARY:
Glucose-6-phosphate dehydrogenase (G6PD) deficiency is prevalent and add a burden on families in Egypt and Middle East due to lifelong diet restriction, non-fava beans diet is main food for most families in the region and parents and doctors consider it as a prohibited food whatever the genetic or clinical phenotypes. The effective management is avoiding a spectrum of food and drugs causing oxidative stress. No data is available about the hazards of consumption of non-fava beans diet.

DETAILED DESCRIPTION:
Investigate the effect of challenge of non-fava beans diet on occurrence of hemolysis in both common and rare mutations causing G6PD deficiency in Egyptian children as well as making a genotype-phenotype correlation. Patients and Methods: The study will include all G6PD deficient children who were regularly followed up in Pediatric Hematology Center, Ain Shams University over last decade from 2004-2014 who stopped eating non fava-bean diet since their diagnosis as G6PD deficient and willing to participate in the diet challenge. They will be enrolled in a one year prospective study involving quantitative analyses for enzymatic activity, and molecular typing of G6PD enzyme using a polymerase chain reaction-amplification refractory mutation system (PCR-ARMS) technique. Patient's medical records will be reviewed as history of blood transfusion and G6PD level at diagnosis. Initial phase will be dietetic challenge with ingestion of non-fava beans taken in small amount (10-20 gm/day for 3 successive days ) for children with haemoglobin level ≥ 11 gm/dl with daily clinical and laboratory monitoring by complete blood count, and markers of hemolysis as well as measurement of malondialdehyde (MDA) level both basal and at study end. A drop of Hb of ≥0.5 gm/dl and / or appearance of hemoglobinuria is considered a significant hemolysis. Patients who will not meet the definition of significant hemolysis will be prospectively followed up for one year with follow up during their chronic exposure by complete blood count and hemolysis markers/ 3 months.

ELIGIBILITY:
Inclusion Criteria:

* All children with proved enzymatic deficiency of G6PD.
* Patients who met the criteria of hemoglobin level at study time ≥ 11 gm/dl

Exclusion Criteria:

* patients with another enzyme deficiency

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Diet challenge | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Hematology clinic, Ain Shams University, Cairo, Egypt